CLINICAL TRIAL: NCT05733481
Title: A Non-Randomized Clinical Study Evaluating Use of the CapBuster System Medical Device for the Crossing of Chronic Total Occlusions in Coronary Arteries
Brief Title: Evaluating the Use of the CapBuster System for the Crossing of CTO's in Coronary Arteries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Praxis Medical Devices Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAP002
Record Dates: First submitted 2023-02-08; First posted 2023-02-17 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Chronic Total Occlusion of Coronary Artery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with the presence of coronary arterial de novo or restenotic chronic total occlusion. (Other): Successful crossing of the targeted chronic total occlusion, defined as angiography confirmed guidewire placement in the true lumen without utilization of a re-entry device.
  Interventions: Device: CapBuster System Medical Device for the Crossing of Chronic Total Occlusions in Coronary Arteries

INTERVENTIONS:
Device: CapBuster System Medical Device for the Crossing of Chronic Total Occlusions in Coronary Arteries — The CapBuster System is a medical device intended to facilitate the intraluminal placement of conventional guidewires beyond chronic total occlusions prior to the utilization of interventional devices. The device system, manufactured by Praxis Medical, comprises the CapBuster support catheter and CapBuster penetrating wire which are mated together with a screw thread.
  Other Names: CapBuster

SUMMARY:
Evaluate the safety and effectiveness of the CapBuster System medical device in crossing de novo or restenotic chronic total occlusions in coronary arteries

DETAILED DESCRIPTION:
Primary Efficacy Endpoints:

Successful crossing of the targeted chronic total occlusion, defined as angiography confirmed guidewire placement in the true lumen without utilization of a re-entry device.

The effectiveness endpoint is designed to demonstrate successful crossing of the chronic total occlusion in at least 80% of lesions.

Primary Safety Endpoints:

Freedom from CapBuster System related clinically significant perforation, embolization, or dissection, defined as perforations or embolization that require intervention and flow-limiting (type C, D, E) dissections.

Secondary Endpoints I. Study procedure success, defined as successful CTO crossing with the absence of in-hospital/outpatient lab significant events and clinically significant perforation, embolization, or dissection not resolved by visual estimate.

II. Evaluation of CTO crossing time. III. Evaluation of total procedural time, fluoroscopic time, and contrast volume.

IV. All CapBuster System related adverse events through 30 days post-procedure. V. Lesion treatment success, defined as ≤ 30% final residual stenosis of the target lesion using commercially available percutaneous treatment modalities.

VI. Freedom from CapBuster System related significant events through 30 days, defined as death or target vessel revascularization that occurred as a result of a CapBuster System related complication or adverse event.

ELIGIBILITY:
Inclusion Criteria:

1. Males > 18 years of age and Female patients of non child-bearing potential
2. Clinical diagnosis of coronary arterial disease requiring revascularization as evidenced by Duplex UltraSound, Digital Subtraction Angiography, CT angiography, or MR angiography
3. Subject requires single- or multi-vessel percutaneous coronary intervention (PCI) of de novo or restenotic target lesion (including in-stent restenotic lesions).
4. Subject's lesion(s) is (are) amenable to stent treatment with currently available CE or FDA-approved stents.
5. Presence of coronary arterial de novo or restenotic chronic total occlusion (100% stenosis), with TIMI 0 flow, confirmed by angiography. Vessel distal to the occlusion(s) must be visualized per collateral or retrograde flow. A maximum of 1 target occlusions can be treated per patient. Target occlusion(s) can be in-stent restenosis
6. Target vessel(s) must be ≥ 2.5 mm and ≤ 3.25 mm in diameter proximal to the target occlusion(s) by visual estimate
7. In the opinion of the investigator, life expectancy of > 1 year
8. Willing and able to sign the informed consent form

Exclusion Criteria:

1. Target occlusion is within a bypass graft
2. acute coronary syndrome with ST elevation,
3. cardiogenic shock or out of hospital cardiac arrest
4. Subject has signs or symptoms of systemic infection/sepsis (temperature ≥38.0o Celsius and WBC ≥12,000 cells/uL). If subject has localized infection, including cellulitis or osteomyelitis, or infection is adequately treated and controlled, per investigator discretion, patient may be enrolled.
5. Known or suspected myocardial infarction or stroke within previous 30 days
6. Currently participating in another investigational drug or device study
7. Female patients of child-bearing potential.
8. Evidence of STEMI within 72 hours of the intended treatment on infarct related or non-infarct related artery.
9. Cardiogenic shock on presentation or during current hospitalization.
10. Known allergies or contraindication to: contrast materials, antiplatelet therapy, aspirin, clopidogrel (Plavix) and ticlopidine (Ticlid), heparin, bivalirudin, stainless steel, or contrast agent (which cannot be adequately premedicated).
11. Subject is currently participating in an investigational drug or device study that has not completed the primary endpoint or that clinically interferes with the current study endpoints. (Note: Trials requiring extended follow-up for products that were investigational, but have since become commercially available, are not considered investigational trials).
12. Stroke or transient ischemic attack within the prior 3 months.
13. Any target vessel that has evidence of excessive thrombus (e.g. requires target vessel thrombectomy).
14. Any target vessel that has evidence of excessive tortuousity (greater than 60 degree angle) that makes it unsuitable for proper stent delivery and deployment,
15. Any target lesion that requires treatment with a device other than percutaneous transluminal coronary angioplasty (PTCA) prior to stent placement (e.g. but not limited to, directional coronary atherectomy, excimer laser, rotational atherectomy, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
CTO crossing of the targeted chronic total occlusion | 30 day follow-up
  Successful crossing of the targeted chronic total occlusion, defined as angiography confirmed guidewire placement in the true lumen without utilization of a re-entry device.
CapBuster System related clinically significant events | 30 day follow-up
  Freedom from CapBuster System related clinically significant perforation, embolization, or dissection, defined as perforations or embolization that require intervention and flow-limiting (type C, D, E) dissections.

SECONDARY OUTCOMES:
Study procedure | 30 day follow-up
  Study procedure success, defined as successful CTO crossing with the absence of in-hospital/outpatient lab significant events and clinically significant perforation, embolization, or dissection caused by use of the CapBuster System

IPD SHARING:
Plan to Share IPD: No
Not intending to share individual patient data